CLINICAL TRIAL: NCT05669391
Title: Randomized Controlled Study on the Effect of Pharmacogenomics on Individualized Precise Treatment of Patients with Depression
Brief Title: Pharmacogenomics on Individualized Precise Treatment of Patients with Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jie Tong, Clinical Professor, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PWZxk2022-18
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2023-01

CONDITIONS: Pharmacogenomics; Depression
Keywords: Pharmacogenomics; depression; Precision treatment; Antidepressants
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacogenomics Group (Experimental)
  Interventions: Diagnostic Test: Genomic analysis of antidepressants
- Non Pharmacogenomics Group (No Intervention)

INTERVENTIONS:
Diagnostic Test: Genomic analysis of antidepressants — Genomic analysis of all antidepressants. Tris EDTA anticoagulation and salting out were used to extract DNA. OD 260/280 was between 1.6-1.8 and the concentration was greater than 50 ng/ μ L。 Using the PCR gene chip detection method and the Asian Screening Array (ASA) chip detection technology of Illumina Company (this chip is the first whole genome SNP chip designed based on the whole genome sequencing data of 9000+East Asian populations, which contains 750000 markers, with 85% of the effective loci), we can obtain the genetic information of polymorphic loci related to the individual differences of drug effects of subjects.
  Arms: Pharmacogenomics Group

SUMMARY:
Based on pharmacogenomics analysis technology, this topic explored its impact on individualized precise treatment of patients with depression through randomized controlled trials. The study subjects were depression patients from the mental health research center affiliated to Tongji University. The sample size was estimated by PASS 21.0.3 software. The sample size of the intervention group and the control group was 60 cases each, and SPSS 25.0 software was used for random sampling. The intervention group completed the pharmacogenomic analysis of antidepressants before using them, and selected appropriate antidepressants according to the characteristics of pharmacokinetics and pharmacodynamics of individual patients, while the control group was administered according to routine treatment. 17 items Hamilton Compression Scale (HAMD-17), Hamilton Anxiety Scale (HAMA), Dimensional Anhedonia Rating Scale (DARS), Pittsburgh sleep quality index (PSQI), Antidepressant Side Effect Checklist (ASEC), Short form 36 item health survey questionnaire (SF-36) (PDQ) assessment. R Project 4.1.1 software was used for statistical analysis of data, PLink v1.07 and Haploview software were used for association analysis of whole genome and drug efficacy and adverse reactions. To explore the difference between the reduction rate of drug efficacy and adverse reactions in patients with depression after pharmacogenomics intervention and conventional treatment. At the same time, we verified and found the gene loci related to the efficacy and adverse reactions of antidepressants in the East Asian population.

ELIGIBILITY:
Inclusion Criteria:

1. Both biological parents are Chinese nationals;
2. Conform to the diagnostic criteria of depression in the fifth edition of the American Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
3. The total score of 17 items of Hamilton Depression Scale (HAMD-17) is ≥ 17;
4. Never used relevant antidepressant drugs;
5. Have a certain visual and auditory discrimination, and have no understanding obstacle;
6. Be able to independently complete the scale measurement;
7. Education level above primary school;
8. Obtain the written informed consent of the patient. If the patient is incapacitated during the onset of the disease, the written informed consent of the legal guardian is required.

Exclusion Criteria:

1. Patients with schizophrenia, schizoaffective disorder, bipolar affective disorder, mental retardation, generalized developmental disorder, delirium, dementia, cognitive dysfunction, alcohol dependence and other diagnoses;
2. Suffering from serious organic diseases, such as diabetes, thyroid disease, hypertension, cardiovascular disease, brain injury, cerebral ischemia or hemorrhage;
3. Patients with narrow angle glaucoma;
4. History of epilepsy and febrile convulsion;
5. Those who have taken drugs in the past;
6. Syphilis specific antibody and AIDS antibody are positive;
7. Those who received MECT or rTMS and other neuromodulation therapy one month before enrollment;
8. The risk assessment indicates that there is a serious suicide attempt or excitement;
9. Laboratory examination indicates that liver function and renal function are impaired;
10. Pregnant or lactating women, or those who plan to have a pregnancy in the near future;
11. Other contraindications of antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Genomic analysis of antidepressants | Baseline
  Using PCR gene chip detection method and Asian Screening Array (ASA) chip detection technology of Illumina Company, we can obtain the genetic information of polymorphic sites related to the individual differences of drug effects of subjects.
17-items Hamilton Depression Scale | Baseline
  Evaluate the severity and treatment effect of the patient's depression within one week.
17-items Hamilton Depression Scale | Week 4
  Evaluate the severity and treatment effect of the patient's depression within one week.
17-items Hamilton Depression Scale | Week 8
  Evaluate the severity and treatment effect of the patient's depression within one week.
17-items Hamilton Depression Scale | Week 16
  Evaluate the severity and treatment effect of the patient's depression within one week.
17-items Hamilton Depression Scale | Week 32
  Evaluate the severity and treatment effect of the patient's depression within one week.
Dimensional Anhedonia Rating Scale | Baseline
  Assess the patient's level of interest, motivation, effort, and happiness in experiencing pleasant activities or experiences.
Dimensional Anhedonia Rating Scale | Week 4
  Assess the patient's level of interest, motivation, effort, and happiness in experiencing pleasant activities or experiences.
Dimensional Anhedonia Rating Scale | Week 8
  Assess the patient's level of interest, motivation, effort, and happiness in experiencing pleasant activities or experiences.
Dimensional Anhedonia Rating Scale | Week 16
  Assess the patient's level of interest, motivation, effort, and happiness in experiencing pleasant activities or experiences.
Dimensional Anhedonia Rating Scale | Week 32
  Assess the patient's level of interest, motivation, effort, and happiness in experiencing pleasant activities or experiences.
Antidepressant Side-Effect Checklist | Baseline
  Evaluate the adverse reactions of patients after using antidepressants.
Antidepressant Side-Effect Checklist | Week 4
  Evaluate the adverse reactions of patients after using antidepressants.
Antidepressant Side-Effect Checklist | Week 8
  Evaluate the adverse reactions of patients after using antidepressants.
Antidepressant Side-Effect Checklist | Week 16
  Evaluate the adverse reactions of patients after using antidepressants.
Antidepressant Side-Effect Checklist | Week 32
  Evaluate the adverse reactions of patients after using antidepressants.
Perceived deficits questionnaire | Baseline
  Assess the patient's subjective cognitive function within one week.
Perceived deficits questionnaire | Week 4
  Assess the patient's subjective cognitive function within one week.
Perceived deficits questionnaire | Week 8
  Assess the patient's subjective cognitive function within one week.
Perceived deficits questionnaire | Week 16
  Assess the patient's subjective cognitive function within one week.
Perceived deficits questionnaire | Week 32
  Assess the patient's subjective cognitive function within one week.

SECONDARY OUTCOMES:
Hamilton Anxiety Scale | Baseline
  Assess the severity of the patient's anxiety symptoms.
Hamilton Anxiety Scale | Week 4
  Assess the severity of the patient's anxiety symptoms.
Hamilton Anxiety Scale | Week 8
  Assess the severity of the patient's anxiety symptoms.
Hamilton Anxiety Scale | Week 16
  Assess the severity of the patient's anxiety symptoms.
Hamilton Anxiety Scale | Week 32
  Assess the severity of the patient's anxiety symptoms.
Pittsburgh sleep quality index | Baseline
  Evaluate the patient's sleep quality within one month, including sleep effect and duration.
Pittsburgh sleep quality index | Week 4
  Evaluate the patient's sleep quality within one month, including sleep effect and duration.
Pittsburgh sleep quality index | Week 8
  Evaluate the patient's sleep quality within one month, including sleep effect and duration.
Pittsburgh sleep quality index | Week 16
  Evaluate the patient's sleep quality within one month, including sleep effect and duration.
Pittsburgh sleep quality index | Week 32
  Evaluate the patient's sleep quality within one month, including sleep effect and duration.
Short-form 36 item health survey questionnaire | Baseline
  Assess the patient's health and quality of life within one month
Short-form 36 item health survey questionnaire | Week 4
  Assess the patient's health and quality of life within one month
Short-form 36 item health survey questionnaire | Week 8
  Assess the patient's health and quality of life within one month
Short-form 36 item health survey questionnaire | Week 16
  Assess the patient's health and quality of life within one month
Short-form 36 item health survey questionnaire | Week 32
  Assess the patient's health and quality of life within one month

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cremonesi L, Carrera P, Cardillo E, Fumagalli A, Lucchiari S, Ferrari M, Righetti SC, Righetti PG, Gelfi C. Optimized detection of DNA point mutations by double gradient denaturing gradient gel electrophoresis. Clin Chem Lab Med. 1998 Dec;36(12):959-61. doi: 10.1515/CCLM.1998.165. PMID 9915229
- [Background] Rush AJ, South C, Jha MK, Jain SB, Trivedi MH. What to Expect When Switching to a Second Antidepressant Medication Following an Ineffective Initial SSRI: A Report From the Randomized Clinical STAR*D Study. J Clin Psychiatry. 2020 Aug 11;81(5):19m12949. doi: 10.4088/JCP.19m12949. PMID 32780949
- [Background] Ahmadimanesh M, Balarastaghi S, Rashedinia M, Yazdian-Robati R. A systematic review on the genotoxic effect of serotonin and norepinephrine reuptake inhibitors (SNRIs) antidepressants. Psychopharmacology (Berl). 2020 Jul;237(7):1909-1915. doi: 10.1007/s00213-020-05550-8. Epub 2020 Jun 11. PMID 32529266
- [Background] Greden JF, Parikh SV, Rothschild AJ, Thase ME, Dunlop BW, DeBattista C, Conway CR, Forester BP, Mondimore FM, Shelton RC, Macaluso M, Li J, Brown K, Gilbert A, Burns L, Jablonski MR, Dechairo B. Impact of pharmacogenomics on clinical outcomes in major depressive disorder in the GUIDED trial: A large, patient- and rater-blinded, randomized, controlled study. J Psychiatr Res. 2019 Apr;111:59-67. doi: 10.1016/j.jpsychires.2019.01.003. Epub 2019 Jan 4. PMID 30677646
- [Background] Hattinger CM, Patrizio MP, Luppi S, Serra M. Pharmacogenomics and Pharmacogenetics in Osteosarcoma: Translational Studies and Clinical Impact. Int J Mol Sci. 2020 Jun 30;21(13):4659. doi: 10.3390/ijms21134659. PMID 32629971
- [Background] Luzum JA, Pakyz RE, Elsey AR, Haidar CE, Peterson JF, Whirl-Carrillo M, Handelman SK, Palmer K, Pulley JM, Beller M, Schildcrout JS, Field JR, Weitzel KW, Cooper-DeHoff RM, Cavallari LH, O'Donnell PH, Altman RB, Pereira N, Ratain MJ, Roden DM, Embi PJ, Sadee W, Klein TE, Johnson JA, Relling MV, Wang L, Weinshilboum RM, Shuldiner AR, Freimuth RR; Pharmacogenomics Research Network Translational Pharmacogenetics Program. The Pharmacogenomics Research Network Translational Pharmacogenetics Program: Outcomes and Metrics of Pharmacogenetic Implementations Across Diverse Healthcare Systems. Clin Pharmacol Ther. 2017 Sep;102(3):502-510. doi: 10.1002/cpt.630. Epub 2017 Jun 9. PMID 28090649
- [Background] Winner JG, Carhart JM, Altar CA, Allen JD, Dechairo BM. A prospective, randomized, double-blind study assessing the clinical impact of integrated pharmacogenomic testing for major depressive disorder. Discov Med. 2013 Nov;16(89):219-27. PMID 24229738
- [Background] Aldrich SL, Poweleit EA, Prows CA, Martin LJ, Strawn JR, Ramsey LB. Influence of CYP2C19 Metabolizer Status on Escitalopram/Citalopram Tolerability and Response in Youth With Anxiety and Depressive Disorders. Front Pharmacol. 2019 Feb 19;10:99. doi: 10.3389/fphar.2019.00099. eCollection 2019. PMID 30837874
- [Background] Gasso P, Rodriguez N, Blazquez A, Monteagudo A, Boloc D, Plana MT, Lafuente A, Lazaro L, Arnaiz JA, Mas S. Epigenetic and genetic variants in the HTR1B gene and clinical improvement in children and adolescents treated with fluoxetine. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Apr 3;75:28-34. doi: 10.1016/j.pnpbp.2016.12.003. Epub 2016 Dec 23. PMID 28025020
- [Background] Health Quality Ontario. Pharmacogenomic Testing for Psychotropic Medication Selection: A Systematic Review of the Assurex GeneSight Psychotropic Test. Ont Health Technol Assess Ser. 2017 Apr 11;17(4):1-39. eCollection 2017. PMID 28515818
- [Derived] Tong J, Yuan J, Qin Y, Zhu N, Zhang T, Zhu X, Xu Y, Liu M, Zhang J, Sun X. Clinicians' experience on the effectiveness of pharmacotherapy in patients with first-episode depression: a randomized controlled trial based on pharmacogenomics. Front Pharmacol. 2025 Aug 7;16:1626654. doi: 10.3389/fphar.2025.1626654. eCollection 2025. PMID 40852613